CLINICAL TRIAL: NCT04040972
Title: Rebalance: Group Compassion Focussed Therapy for People With Transdiagnostic Chronic Health Conditions - a Case Series
Brief Title: Rebalance: Compassion Focused Therapy in a Transdiagnostic Health Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/SS/0164
Record Dates: First submitted 2019-07-23; First posted 2019-08-01 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Psychological Adjustment; Compassion; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rebalance - Group Compassion Focussed Therapy (Experimental)
  Interventions: Other: Compassion Focussed Therapy

INTERVENTIONS:
Other: Compassion Focussed Therapy — Group compassion focussed therapy. One session every week for 10 weeks. Each session lasts 2.5 hours with two breaks during this time.

SUMMARY:
This study evaluates the use of group Compassion Focussed Therapy in a population with various and/or multiple long term health conditions. A multiple baseline, single case experimental design will be used with a view to evaluate changes in psychological adjustment and compassion. Daily data and weekly questionnaire batteries will be collected across a baseline period and ten weeks of group intervention. Participants will be those already referred to the group by a clinician as part of their routine care.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing difficulties adjusting to one or more chronic physical health condition(s)
* Willing and motivated to attend a nine-week group facilitated in English
* Exhibit sufficient interpersonal skills and impulse control to allow them to engage with group members without disrupting group dynamics
* Able to provide informed consent

Exclusion Criteria:

* Moderate or severe impairment of cognitive function
* Primary problem related to drug or alcohol misuse
* Actively suicidal or experiencing an acute deterioration in their mental health including experiencing an acute psychotic episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
The compassionate engagement and action scales (assessing change over time) | Recorded weekly throughout baseline period and ten week intervention. Also collected once at 3 month follow up.
  Measure of compassion compromising three subscales. Each scale contains two sub-sections. All answers on scale of 1 (Never) to 10 (Always).
Work and social adjustment scale (assessing change over time) | Recorded weekly throughout baseline period and ten week intervention. Also collected once at 3 month follow up
  A 5-item measure of functional impairment due to a specified stressor. Each question is scored 1 (Not at all) to 8 (very severely)
Self-efficacy for managing chronic disease scale (assessing change over time) | Recorded weekly throughout baseline period and ten week intervention. Also collected once at 3 month follow up
  A 6-item measure of perceived self-efficacy to adherence to recommended self-management programs. Each item scored 1 (not at all confident) to 10 (totally confident).
Illness Cognition Questionnaire (assessing change over time) | Recorded weekly throughout baseline period and ten week intervention. Also collected once at 3 month follow up
  18 items each rated on a four-point scale with high internal validity (all above 0.81. Assessing three domains of perceiving illness (helplessness, acceptance and perceived benefits) this tool identifies maladaptive cognitive styles surrounding illness which are linked to poorer psychological outcomes. Scored 1 (not at all) to 4 (completely)
The Warwick-Edinburgh Mental Well-being scale (assessing change over time) | Recorded weekly throughout baseline period and ten week intervention. Also collected once at 3 month follow up
  A 14 item measure of psychological wellbeing scored 1 (none of the time) to 5 (all of the time).

SECONDARY OUTCOMES:
Daily diary questions (assessing change over time) | Daily throughout baseline (14-5 days) and intervention (10 weeks). May also be collected for 7 days at time of three month follow up.
  3 questions relating to the participants sense of adjustment and self-compassion on that day. Each question uses a five-point likert scale from 1 (very poorly) to 5 (very well)

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian Clinical Health Psychology Service, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No